CLINICAL TRIAL: NCT03960229
Title: The Evaluation of the Effect of Microfluidic Sperm Sorting Chip 'Labs-on-a-chip' on IVF Success in Male Factor: a Randomized Controlled Trial
Brief Title: The Evaluation of the Effect of Microfluidic Sperm Sorting Chip 'Labs-on-a-chip' on IVF Success in Male Factor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Yeditepe University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BezmialemVU microchip study
Record Dates: First submitted 2018-12-05; First posted 2019-05-23 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Male Infertility; Infertility, Male
Keywords: microfluid chip; gradient-density; IVF; male factor
MeSH Terms: conditions — Infertility, Male | interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MicroFluidic Sperm Sorting Chips (Experimental): Sperm Sorting microfluidic chips (for ICSI) will be used when preparing sperm of male partner and microinjection (ICSI) will be made with separated sperm
  Interventions: Other: MicroFluidic Sperm Sorting Chips
- gradient-density centrifugation (Active Comparator): gradient-density centrifugation technique will be used when preparing sperm of male partner and microinjection (ICSI) will be made with separated sperm
  Interventions: Other: Gradient-Density Centrifugation

INTERVENTIONS:
Other: MicroFluidic Sperm Sorting Chips — sperm selection of IVF treatment
  Arms: MicroFluidic Sperm Sorting Chips
Other: Gradient-Density Centrifugation — sperm selection of IVF treatment
  Arms: gradient-density centrifugation

SUMMARY:
Microfluidic chips are one of the methods of sperm separation to eliminate DNA fragmentation in sperm. It is thought that the separation of sperm by centrifugation in the classical gradient density (Percoll) method used in sperm separation in IVF (in vitro fertilization) laboratories leads to the increase of reactive oxygen radicals in sperm and this leads to sperm DNA fragmentation. Studies comparing Percoll and microfluidic chip method in terms of sperm, embryo quality and pregnancy rates are limited. In this context, it is aimed to investigate the effect of Percoll or Microfluidic Chip Technology on the quality of sperms and embryos obtained with these sperms and their pregnancy rates prospectively.

DETAILED DESCRIPTION:
The increase in male infertility rate due to environmental and physiological conditions leads to an increase in the use of assisted reproductive techniques. Isolation of living and morphologically normal live sperm is an integrated procedure in commonly used IVF / ICSI(intracytoplasmic sperm injection) / IUI(intrauterine insemination) procedures. Although current IVF / ICSI procedures result in a successful pregnancy of around 50%, the process can be greatly compromised if the selected sperm is abnormal. Microfluidic chips are one of the recommended sperm separation methods to eliminate DNA fragmentation in sperm. It is thought that the separation of the sperm by centrifugation in the classical gradient density (Percoll) method which is used in the separation of sperm in the IVF Laboratories, causes the increase of reactive oxygen radicals in sperm and this leads to sperm DNA fragmentation. Studies comparing Percoll and microfluidic chip method in terms of sperm, embryo quality and pregnancy rates are limited. In this context, it is aimed to investigate the effect of Percoll or Microfluidic Chip Technology on the quality of sperms and embryos obtained with these sperms and their pregnancy rates prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Apply to the IVF clinic due to male factor
* Volunteer

Exclusion Criteria:

* Inadequate follicle development with medication
* Embryo does not have the appropriate quality for transfer
* Female-induced infertility
* Refuse to participate in research

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 139 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Compare microfluid chip and density-gradient methods in terms of IVF success | average of 1 year
  measure the clinical pregnancy rate by using serum beta-HCG (human chorionic gonadotropin) level.
Compare microfluid chip and density-gradient methods in terms of embryo quality | average of 1 year
  Embryo morphology will be assessed on day 3 using the standard criteria of the number of blastomeres and extent of fragmentation and blastomere asymmetry. Top quality embryos on day 3 will be designated as embryos with 7-8 cells, ≤10% fragmentation, and symmetric blastomeres. Using these criteria, the rate of top quality embryos will be analyzed.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bezmialem University, Istanbul
  - Yeditepe University, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asghar W, Velasco V, Kingsley JL, Shoukat MS, Shafiee H, Anchan RM, Mutter GL, Tuzel E, Demirci U. Selection of functional human sperm with higher DNA integrity and fewer reactive oxygen species. Adv Healthc Mater. 2014 Oct;3(10):1671-9. doi: 10.1002/adhm.201400058. Epub 2014 Apr 17. PMID 24753434
- [Background] Tasoglu S, Safaee H, Zhang X, Kingsley JL, Catalano PN, Gurkan UA, Nureddin A, Kayaalp E, Anchan RM, Maas RL, Tuzel E, Demirci U. Exhaustion of racing sperm in nature-mimicking microfluidic channels during sorting. Small. 2013 Oct 25;9(20):3374-84. doi: 10.1002/smll.201300020. Epub 2013 May 16. PMID 23677651
- [Background] Nosrati R, Graham PJ, Zhang B, Riordon J, Lagunov A, Hannam TG, Escobedo C, Jarvi K, Sinton D. Microfluidics for sperm analysis and selection. Nat Rev Urol. 2017 Dec;14(12):707-730. doi: 10.1038/nrurol.2017.175. Epub 2017 Oct 31. PMID 29089604